Date: 11/15/2023

National Clinical Trials #: NCT05803720

Study Title: Development of an Online Provider Intervention to Address Intersectional Stigma and Medical Mistrust in People Living with HIV

#### **HIV Care Provider Training to Address Medical Mistrust**

#### **VERBAL AGREEMENTS TO PARTICIPATE**

We are inviting you to participate in this research study that is developing an online provider training to address stigma and medical mistrust. Your participation throughout the study is completely voluntary. You should feel free to ask any questions and should understand the study completely before you agree to participate.

### Who is doing the study?

Investigators from the RAND Corporation, California Prevention Training Center, and Brigham & Women's Hospital are conducting the study. The National Institutes of Mental Health provides funding for this study.

#### What is the goal of this study?

The goal of this study is to develop and pilot test a provider training for HIV care providers to understand and address the impact of stigma and medical mistrust. We are recruiting about 10 HIV care providers.

## Who can participate in this study?

You are eligible to participate if you meet the following criteria:

- An HIV health care provider, providing care for people at risk for or living with HIV
- Working primarily with Black and Latino/a/x patients or clients
- Can make the time commitment to participate in the study (i.e., attending the training for up to 4 hours and provide qualitative feedback)

## What will we ask you to do?

If you are eligible and decide to participate, you will be asked to do the following:

- 1. Participate in an online training: You will be asked to participate in a provider training session (up to 4 hours) via remote web-based platforms to learn about stigma and medical mistrust commonly experienced by Black and Latino/a/x patients or clients. The virtual training may be offered in one setting or on two separate days. The training session will be audio-recorded so that we can monitor how well the trainers are conducting the training and make refinement to training material. The training involves didactic, educational information and skill training contents (e.g., learning new skills through demonstration, discussion, and role play).
- 2. Interview: After completing the training, we will also ask you to complete an interview with one of our research staff. The interview will ask your qualitative feedback about the acceptability of the training program, such as how you feel about the training, what suggestions you may have about improving the training, and other topics. Your feedback will be used to improve the training before we test it in a larger group of providers.

#### What are the potential benefits of participating?

There is no cost for participating in this study. We hope you may find the provider training materials helpful and can potentially increase your competence for understanding and addressing stigma and medical mistrust related issues in your clinical work.

### What are the potential risks of participating?

There are no physical risks to participate in this study and we anticipate minimal psychological risks. The provider training and interview will involve asking questions and eliciting discussion within your professional capacity.

## How is confidentiality protected?

All the information that you provide to us will be kept private and confidential, and only trained and designated research staff will have access to the information, including personal information that would identify you. During the consent procedure, we will obtain your personal contact information, including your name, email address (required), and phone number. The personal contact information will only be used to send you incentives.

For providers who are selected to take part in the provider training and interview, these sessions and interviews will be audio-recorded. We will ask participants not to use any names on these recordings that may identify specific individuals; we will remove all reference to names or other identifiers from interview transcripts. We will also destroy all recordings at the end of the study.

To help us protect your privacy further, we have a federal Certificate of Confidentiality. This certificate assures that the RAND Corporation and their staff may not be forced to identify you in any civil, criminal, administrative, legislative, or other proceedings, whether state, federal, or local. The exception is if keeping specific information private would immediately put you in danger, or put in danger someone else we know about (such as if you tell us about child or elder abuse).

De-identified data from this study may be shared with other researchers. To de-identify your data, all personal information such as name and phone number will be removed and replaced with a code number. Other researchers can then file an application with this study's Principal Investigator, Dr. Lu Dong, to obtain access to your de-identified study data for research purposes. The Principal Investigator and members of RAND's Human Subjects Protections Committee, who know how to protect health and science information, will look at every request carefully to minimize risks to your privacy. By sharing data, researchers hope to learn new and important things about HIV care more quickly than before. If you do not want your data to be shared with other researchers, you may contact the Principal Investigator, Dr. Dong.

### What incentives will you receive for participating in the study?

You will receive \$150 for completing the training and an additional \$50 for completing the interview at the end of the training.

## Who to contact if you have questions about the study?

If you have questions about the study before you make the decision to participate, or if you have any concerns after you decide to participate, please contact the main study investigator: Dr. Lu Dong at RAND, 1776 Main Street, Santa Monica, CA, 90407, email: <a href="mailto:ldong@rand.org">ldong@rand.org</a>, phone: 1-800-447-2631 x7494.

If you have questions about your rights as a research participant or need to report a research-related injury or concern, you can contact RAND's Human Subjects Protection Committee toll-free at (866) 697-5620 or by emailing <a href="mailto:hspcinfo@rand.org">hspcinfo@rand.org</a>. When you contact the Committee, please reference Project #2021-N0035.

#### Consent

#### **Participant Statement:**

- I have read this consent form
- I understand the information this consent form provides
- I willingly agree to take part in this research study
- I have been provided with a copy of this consent form
- I agree to allow the research team to contact me about future research study conducted by the team

### Authorization to Record

## What am I being asked to Authorize?

RAND would like to record portions of the provider training sessions in which you will be participating and use the video and audio recording it creates for the following purposes:

Modifying and refining the training materials for future use

# How will the recording be used by RAND?

The recording will be used solely for the purposes identified in this document. The RAND research team will not use the recording for any other purpose without your approval. RAND intends to make the recording available to members of the research team involved in modifying and refining the training materials but will not distribute them beyond this purpose. You will not be identified by name in any video or audio recording.

The recordings may be used by the RAND research team only until 04/30/2025.

### Release Authorization

By providing verbal consent, which will be videorecorded, I authorize the research team at the RAND Corporation ("RAND") to use this recording for the purposes identified above.

Additionally, I understand and agree that:

- I will not receive any payment for my appearance in, or RAND's use of, any video or audio recording.
- I am waiving any and all commercial and publicity rights that I may have (or my family or heirs may have) with respect to the video and/or audio recording.
- There are no limitations on how the video or audio recordings will be used except as stated in this
  document.

I am eighteen years of age or older (or an emancipated minor) and, to the best of my knowledge, am legally capable of entering into agreements in my own name.